CLINICAL TRIAL: NCT06432322
Title: Effects of Esketamine Challenge on Brain Glutamate Release (fMRS), Resting State Connectivity (BOLD-rs-fMRI), and Neuroplasticity (Visual Task)
Brief Title: (GluEsk) Glutamate and Esketamine
Acronym: GluEsk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R90468/RE001
Record Dates: First submitted 2024-05-21; First posted 2024-05-29 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: Esketamine; Brain glutamate release; fMRS; Resting state connectivity; BOLD-rs-fMRI; Neuroplasticity; Visual task; Healthy volunteers; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Within-subject, cross-over design
Who Masked: Participant, Outcomes Assessor
Masking Description: Self-administered by the participant wearing an eye mask, following instructions and under supervision of appropriately trained medical staff where resuscitation facilities are available, via a single-use device delivering 28 mg as two sprays (i.e., one spray per nostril).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esketamine (Experimental): Nasal spray solution, 56mg (28mg per nostril), intranasal
  Interventions: Drug: Esketamine nasal spray
- Placebo (Placebo Comparator): Nasal spray solution, 0.9% NaCl, intranasal
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Esketamine nasal spray — Nasal spray solution, 56mg (28mg per nostril), intranasal
  Arms: Esketamine
Other: Placebo — Nasal spray solution, 0.9% NaCl, intranasal
  Arms: Placebo

SUMMARY:
Esketamine is the S-enantiomer of racemic ketamine, a N-methyl-D-aspartate (NMDA) receptor antagonist. Esketamine and other antidepressant NMDA receptor antagonists are hypothesised to act by producing a rapid increase in brain glutamate release, which then stimulates α-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA) receptors. This activity in turn is thought to restore synaptic functioning, neuroplasticity, and connectivity in brain regions involved in mood regulation, which would be ultimately responsible for the antidepressant effect of esketamine. However, the effect of esketamine on glutamate release in humans has not previously been studied. In this study we therefore aim to ascertain the effect of esketamine on dynamic brain glutamate release, resting state connectivity, and neuroplasticity as measured via fMRS, BOLD-rs-fMRI, and a behavioural computerised visual task respectively.

DETAILED DESCRIPTION:
There is growing interest in the use of antagonists at the glutamate N-methyl-D-aspartate (NMDA) receptor in patients with treatment-resistant depression (TRD). Work in animal studies suggests that NMDA receptor antagonists act initially by increasing brain glutamate release, but whether such an action occurs in humans is not established.

Esketamine is the S-enantiomer of racemic ketamine: a non-selective, non-competitive, antagonist of the ionotropic glutamate NMDA receptor. It is the only NMDA receptor antagonist licensed in the UK for the treatment of patients with TRD. Esketamine is administered intranasally: it is rapidly absorbed by the nasal mucosa following nasal administration and can be measured in plasma within 7 minutes following a 28 mg dose. The time to reach maximum plasma concentration (tmax) is typically 20 to 40 minutes after the last nasal spray of a treatment session. It is hypothesised that through NMDA receptor antagonism, esketamine produces a transient increase in glutamate release leading to increases in α-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA) receptor stimulation and subsequently to increases in neurotrophic signalling which may contribute to the restoration of synaptic function, neuroplasticity, and connectivity in brain regions involved with the regulation of mood.

Glutamate is the primary excitatory neurotransmitter in the brain and has been implicated in several neuropsychiatric disorders. "Gold-standard" methods to assess glutamate activity in the living human brain are expensive and involve radioactive injections and invasive blood sampling. More recently, preliminary work in our Clinical Psychopharmacology laboratory (Department of Psychiatry, University of Oxford) has shown that 7T fMRS (a more widely available, non-invasive, safe technique) that uses a visual stimulus ("flickering checkerboard") can reliably and sensitively measure changes in brain glutamate release. No prior study however has shown whether this effect is susceptible to pharmacological challenge. We therefore propose to assess whether through its NMDA/AMPA-mediated activity, esketamine induced glutamate increase can be measured via this fMRS technique.

The aims of this study are to investigate the effect of esketamine on brain glutamate release and resting state connectivity, and on vision. Therefore, the primary objective of this study is to assess the effect of a single dose of esketamine 56mg intranasal vs placebo on brain glutamate release changes measured via 7T fMRS "flickering checkerboard" stimulus. Secondary objectives include the investigation of the effects of esketamine on brain resting state connectivity changes measured via 7T BOLD-rs-fMRI, and on vision measured via a behavioural computerised visual task. Psychological questionnaires will also be measured to check for possible correlations with the outcomes measured.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years
* Body Mass Index in the range of 18-30
* Sufficiently fluent in English to understand the study instructions
* Willing and able to give informed consent for participation in the research

Exclusion Criteria:

* Currently on any regular prescribed medications (except the contraceptive pill), unless unlikely to compromise safety or affect data quality in the opinion of the Investigator
* Known hypersensitivity to the study drug (i.e., esketamine)
* History of, or current significant alcohol or substance misuse disorder
* Any use of recreational drugs over the last 3 months
* Any lifetime use of ketamine or phencyclidine (PCP)
* Currently smoking >/=20 cigarettes/day
* History of, or current significant cardiovascular disorder (e.g., hypertension, myocardial infarction)
* History of, or current significant neurological disorder (e.g., epilepsy, migraine) or cerebrovascular disorder (e.g., haemorrhagic or ischemic stroke, aneurysmal vascular disease, raised intracranial pressure)
* History of, or current significant respiratory, hepatic, urinary tract, or thyroid disorders
* History of, or current acute porphyria
* History of, or current significant psychiatric disorder (e.g., psychosis, mania, depression)
* History of, or current eye disorder, not including refractive error that can be corrected with glasses or contact lenses)
* Pregnant, breast feeding, women of child-bearing potential not using appropriate contraceptive measures
* Any contraindication to 7T MRI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Brain Glutamate Dynamic Change | Acute (40-60 minutes after nasal spray application)
  From the functional magnetic resonance spectroscopy (fMRS), calculating the glutamate concentration change in response to flickering checkerboard stimulation (by the difference in the rest concentrations to the stimulation concentrations). This dynamic glutamate change will be compared between individuals on ketamine and placebo, in a within subject cross over design.

SECONDARY OUTCOMES:
Brain Glutamate Baseline Change | Acute (40-60 minutes after nasal spray application)
  Determining if the baseline glutamate concentration levels in the rest condition is different between individuals on ketamine and placebo (without the influence of a functional task to produce a dynamic change).
Excitatory-Inhibitory Ratio Change | Acute (40-60 minutes after nasal spray application)
  Using the glutamate and GABA concentrations quantified from the fMRS data, we will calculate the glu-GABA ratio to assess the excitatory-inhibitory ratio, and determine whether this ratio is different between the ketamine and placebo conditions.
Brain Resting State Connectivity | Acute (40-60 minutes after nasal spray application)
  Brain resting state connectivity change measured via blood oxygenation level-dependent resting-state functional Magnetic Resonance Imaging (BOLD-rs-fMRI) 7T, comparing ketamine and placebo conditions.
Visual response | Post-Acute (60-120 minutes after nasal spray application)
  Behavioural visual response measured via a computerised visual task, in both the ketamine and placebo conditions we will be comparing differences in the binocular rivalry perceptual suppression, differences in orientation discrimination thresholds and differences in stereopsis thresholds.
Exploratory Analysis of Other Metabolite Concentrations at Baseline or Changes After Stimulation | Acute (40-60 minutes after nasal spray application)
  Other metabolites captured from the fMRS STEAM sequence will be analysed to assess whether there are differences between the concentrations in the ketamine and placebo conditions, whether that be dynamic or baseline concentration changes.
Exploratory Investigation of the Influence of Age, Gender, and Questionnaire Scores on Metabolite Concentration Change | Acute (40-60 minutes after nasal spray application)
  Data collected on demographic factors like age and sex and questionnaire scores will be assessed to determine if they significantly influence metabolite levels.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo De Giorgi, MD, DPhil, MRCPsych, Principal Investigator — University of Oxford, Department of Psychiatry
Locations (1):
- Department of Psychiatry, University of Oxford, Warneford Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ip IB, Berrington A, Hess AT, Parker AJ, Emir UE, Bridge H. Combined fMRI-MRS acquires simultaneous glutamate and BOLD-fMRI signals in the human brain. Neuroimage. 2017 Jul 15;155:113-119. doi: 10.1016/j.neuroimage.2017.04.030. Epub 2017 Apr 19. PMID 28433623
- [Background] Jewett BE, Thapa B. Physiology, NMDA Receptor. 2022 Dec 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK519495/ PMID 30137779
- [Background] Li CT, Yang KC, Lin WC. Glutamatergic Dysfunction and Glutamatergic Compounds for Major Psychiatric Disorders: Evidence From Clinical Neuroimaging Studies. Front Psychiatry. 2019 Jan 24;9:767. doi: 10.3389/fpsyt.2018.00767. eCollection 2018. PMID 30733690
- [Background] Rosenbaum SB, Gupta V, Patel P, Palacios JL. Ketamine. 2024 Jan 30. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470357/ PMID 29262083